CLINICAL TRIAL: NCT05135780
Title: Phase Project (Fundació Albert Salut i Educació): Effects of a Multidisciplinary Intervention (Osteopathy and Social Work) on the Quality of Life in Children at Social Risk. A Case Series Protocol
Brief Title: The Quality of Life in Children at Social Risk, a Case Series Study Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Francesco Cerritelli (Other)
Collaborators: Come Collaboration (Other); Fundació Albert Salut i Educació (Unknown)
Responsible Party: Sponsor-Investigator, Francesco Cerritelli, President of Come Collaboration, Come Collaboration
Organization: Come Collaboration (Other)
Other Study IDs: 26102021
Record Dates: First submitted 2021-10-26; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Osteopathic Medicine; Effectiveness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Osteopathic manual treatment — Between 5 and 8 sessions of osteopathy will be carried out, and the time interval between sessions may vary depending on the need and individual evolution of each child, assessed by the team of osteopaths.
Other: Social education — * Intervention in children:
    * During the school year there will be activities of two days per week with a duration of 2.5 hours per session in the afternoon.
    * The activities will focus on school reinforcement, facilitating snacks and having a recreational space.
    * Groups will be made by age ranges (from 4 to 6 and from 7 to 12) of maximum 10 children, due to the current COVID situation. The number could vary in the event of a change in measures at the institutional level.
  * Family intervention:
    * Quarterly tutoring spaces between the coordinators and the team of social educators to evaluate needs, specify objectives and assess evolution.
    * Monthly group spaces for mothers managed by the team of educators where they will exchange experiences and create an informal support network.
    * Monthly spaces shared between parents and children accompanied by the educational team, where family ties will be worked through play.

SUMMARY:
this case series study has the aim to observe the effect of a multidisciplinary intervention (social accompaniment, school reinforcement and osteopathic treatment) on the quality of life of children with social risk in primary school age.

DETAILED DESCRIPTION:
To observe the effect of a multidisciplinary intervention (social accompaniment, school reinforcement and osteopathic treatment) on the quality of life of children with social risk in primary school age.

II. Secondary objectives

* Observe if the quality of life of children in whom an osteopathic intervention is performed to the family, improves in relation to children who are not treated to the family.
* Observe if the number of sessions has any impact on the evolution of the quality of life of children.
* Observe whether age is an influential factor for improving children's quality of life.
* Observe the possible confounding factors that may influence the evolution of children's quality of life. These factors are detailed later in the section on secondary variables.
* Observe if there is a decrease in pain, in children who refer it.
* Observe if there is an improvement in the different reasons for consultation.

  * The coordination of the study and its different interventions will be carried out from the AF. Carrer Consolat de Mar, 45. Barcelona.
  * Osteopathic intervention will be performed in AF. It is decided to move the Solidarity Osteopathy Service to the AF, outside the FOB Osteopathy Clinic, to bring the solidarity service closer to a more appropriate and closer district for the patient at social risk. Having to move outside their environment, taking public transport, language problems and comparative grievances with the utilitarians of a private service turned out to be reasons for absenteeism and lack of commitment. The transfer has been a success and we believe it is convenient to carry out the study within the FA to preserve the location of the project and the comfort/safety of users at social risk.
  * The participating families will be referred, as is usually worked in this foundation, by the Social Services Centers, other agents and social entities, CSMIJ (Center for Mental Health of Children and Youth), CDIAP (Center for Development and Early Care), EAIA (Child and Adolescent Care Teams), public schools in the Ciutat Vella district of the city of Barcelona (Cervantes, Angel Baixeras, Parc de la Ciutadella, Alexandre Galí, Pere Vila), or families who have requested assistance directly.
  * The Covid protocol that is in force during the start of the study will be taken into account.
  * The coordination of the study and its different interventions will be carried out from the AF. Carrer Consolat de Mar, 45. Barcelona.
  * Osteopathic intervention will be performed in AF. It is decided to move the Solidarity Osteopathy Service to the AF, outside the FOB Osteopathy Clinic, to bring the solidarity service closer to a more appropriate and closer district for the patient at social risk. Having to move outside their environment, taking public transport, language problems and comparative grievances with the utilitarians of a private service turned out to be reasons for absenteeism and lack of commitment. The transfer has been a success and we believe it is convenient to carry out the study within the FA to preserve the location of the project and the comfort/safety of users at social risk.
  * The participating families will be referred, as is usually worked in this foundation, by the Social Services Centers, other agents and social entities, CSMIJ (Center for Mental Health of Children and Youth), CDIAP (Center for Development and Early Care), EAIA (Child and Adolescent Care Teams), public schools in the Ciutat Vella district of the city of Barcelona (Cervantes, Angel Baixeras, Parc de la Ciutadella, Alexandre Galí, Pere Vila), or families who have requested assistance directly.
  * The Covid protocol that is in force during the start of the study will be taken into account.
  * The coordination of the study and its different interventions will be carried out from the AF. Carrer Consolat de Mar, 45. Barcelona.
  * Osteopathic intervention will be performed in AF. It is decided to move the Solidarity Osteopathy Service to the AF, outside the FOB Osteopathy Clinic, to bring the solidarity service closer to a more appropriate and closer district for the patient at social risk. Having to move outside their environment, taking public transport, language problems and comparative grievances with the utilitarians of a private service turned out to be reasons for absenteeism and lack of commitment. The transfer has been a success and we believe it is convenient to carry out the study within the FA to preserve the location of the project and the comfort/safety of users at social risk.
  * The participating families will be referred, as is usually worked in this foundation, by the Social Services Centers, other agents and social entities, CSMIJ (Center for Mental Health of Children and Youth), CDIAP (Center for Development and Early Care), EAIA (Child and Adolescent Care Teams), public schools in the Ciutat Vella district of the city of Barcelona (Cervantes, Angel Baixeras, Parc de la Ciutadella, Alexandre Galí, Pere Vila), or families who have requested assistance directly.
  * The Covid protocol that is in force during the start of the study will be taken into account.
  * The coordination of the study and its different interventions will be carried out from the AF. Carrer Consolat de Mar, 45. Barcelona.
  * Osteopathic intervention will be performed in AF. It is decided to move the Solidarity Osteopathy Service to the AF, outside the FOB Osteopathy Clinic, to bring the solidarity service closer to a more appropriate and closer district for the patient at social risk. Having to move outside their environment, taking public transport, language problems and comparative grievances with the utilitarians of a private service turned out to be reasons for absenteeism and lack of commitment. The transfer has been a success and we believe it is convenient to carry out the study within the FA to preserve the location of the project and the comfort/safety of users at social risk.
  * The participating families will be referred, as is usually worked in this foundation, by the Social Services Centers, other agents and social entities, CSMIJ (Center for Mental Health of Children and Youth), CDIAP (Center for Development and Early Care), EAIA (Child and Adolescent Care Teams), public schools in the Ciutat Vella district of the city of Barcelona (Cervantes, Angel Baixeras, Parc de la Ciutadella, Alexandre Galí, Pere Vila), or families who have requested assistance directly.
  * The Covid protocol that is in force during the start of the study will be taken into account.
  * The coordination of the study and its different interventions will be carried out from the AF. Carrer Consolat de Mar, 45. Barcelona.
  * Osteopathic intervention will be performed in AF. It is decided to move the Solidarity Osteopathy Service to the AF, outside the FOB Osteopathy Clinic, to bring the solidarity service closer to a more appropriate and closer district for the patient at social risk. Having to move outside their environment, taking public transport, language problems and comparative grievances with the utilitarians of a private service turned out to be reasons for absenteeism and lack of commitment. The transfer has been a success and we believe it is convenient to carry out the study within the FA to preserve the location of the project and the comfort/safety of users at social risk.
  * The participating families will be referred, as is usually worked in this foundation, by the Social Services Centers, other agents and social entities, CSMIJ (Center for Mental Health of Children and Youth), CDIAP (Center for Development and Early Care), EAIA (Child and Adolescent Care Teams), public schools in the Ciutat Vella district of the city of Barcelona (Cervantes, Angel Baixeras, Parc de la Ciutadella, Alexandre Galí, Pere Vila), or families who have requested assistance directly.
  * The Covid protocol that is in force during the start of the study will be taken into account.

ELIGIBILITY:
Inclusion Criteria:

* The children will be selected from the set of users of the Albert Foundation with the following criteria:

  * Children from families at social risk, in school and aged between 6 and 12 years of age. The situation of social risk or vulnerability will be determined by the "Instrument de cribratge de les situacions de risc i de desemparament" of the General Directorate of Child Care (DGAIA) of the Generalitat de Catalunya (41), being referred by Social Services, other social entities or that have requested assistance directly.

Exclusion Criteria:

* ○ Families who do not sign consent to participate in the study.

  * The unavailability of families to participate in the study. In some cases, even if there are children who meet the inclusion criteria, they may not have the capacity to participate for reasons outside the AF or/or personal.

Ages: 6 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: * The participating families will be referred, as is usually worked in this foundation, by the Social Services Centers, other agents and social entities, CSMIJ (Center for Mental Health of Children and Youth), CDIAP (Center for Development and Early Care), EAIA (Child and Adolescent Care Teams), public schools in the Ciutat Vella district of the city of Barcelona (Cervantes, Angel Baixeras, Parc de la Ciutadella, Alexandre Galí, Pere Vila), or families who have requested assistance directly.
  * The Covid protocol that is in force during the start of the study will be taken into account
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Quality of Life Inventory (PedsQL) questionnaire | -1rst questionnaire at baseline 2nd questionnaire in December 2021. - 3rd questionnaire in March 2022. - 4th questionnaire in June 2022.
  The PedsQL is a brief, standardized, generic assessment instrument that systematically assesses patients' and parents' perceptions of self-report of health-related quality of life in pediatric patients with chronic health conditions. Is a 23-item generic health status instrument. Items are scored from 5-point Likert scale from 0 (Never) to 4 (Almost always) Scores then are transformed on a scale from 0 to 100. Step 1: Transform Score
  Items are reversed scored and linearly transformed to a 0-100 scale as follows:
  0=100, 1=75, 2=50, 3=25, 4=0. Mean score = Sum of the items over the number of items answered. If 50% or more items are completed: Impute the mean of the completed items in a scale.

SECONDARY OUTCOMES:
Number of Osteopathy sessions | july 2022
  Number of osteopathy sessions needed for each child and/or family.
Change in Numerical Pain Scale | At baseline and second measure at July 2022
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Roura Carvajal, MsC, Study Director — Sonia
Locations (1):
- Sonia Roura Carvajal, La Seu d'Urgell, Spain

IPD SHARING:
Plan to Share IPD: Undecided